CLINICAL TRIAL: NCT05421234
Title: Effect of COVID-19 on Spermiogram, Platelet Mitochondrial Bioenergetic, Antioxidants and Oxidative Stress in Infertile Men
Brief Title: Effect of COVID-19 on Platelet Mitochondrial Bioenergetic, Antioxidants and Oxidative Stress in Infertile Men.
Acronym: COVInfertility
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Comenius University (Other)
Collaborators: GYN-FIV (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: COVID-19-INFERTILITY-SK01/2022
Record Dates: First submitted 2022-06-15; First posted 2022-06-16 (Actual); Last update posted 2022-06-22 (Actual); Status verified 2022-01

CONDITIONS: Infertility, Male; COVID-19
Keywords: men infertility; after-COVID-19; platelets; mitochondrial bioenergetics; coenzyme Q10; oxidative stress
MeSH Terms: conditions — Infertility, Male; COVID-19

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- infertile men with post-COVID-19 (vaccinated or without vaccination) (Active Comparator): 15 infertile men with post-COVID-19 (vaccinated or without vaccination)
  Interventions: Other: diagnostic test and sperm analysis
- infertile men without post-COVID-19 (vaccinated or without vaccination) (Active Comparator): 15 infertile men without post-COVID-19 (vaccinated or without vaccination)
  Interventions: Other: diagnostic test and sperm analysis
- Control: 15 healthy men volunteers (no COVID-19, no other pathologies) (Active Comparator): 15 healthy men volunteers (no COVID-19, no other pathologies) as control group
  Interventions: Other: diagnostic test and sperm analysis

INTERVENTIONS:
Other: diagnostic test and sperm analysis — Diagnostic Test: 2x14 ml of peripheral blood collected in the tube with anticoagulant, for platelet isolation, respirometry mitochondrial analysis, antioxidants (coenzyme Q10, vitamin E, gamma-tocopherol, beta-carotene) and TBARS estimation.
  Sperm analysis: standard spermiogram examination (volume, pH, number, motility and pathology) in the broker chamber, as well as extended examinations: mioxsys for redox potential, Vitalsperm (eosin-nigrosine staining) for sperm vitality and anti-sperm antibody (IgG) test.

SUMMARY:
To verify the hypothesis that infertility and the effect of SARS-CoV-2 on infertility may damage platelet mitochondrial bioenergetics and endogenous coenzyme Q10 levels in infertile men.

DETAILED DESCRIPTION:
Infertility is defined as the failure of the reproductive system to achieve pregnancy after 12 months of unprotected sex life. The pathobiochemical mechanisms of male fertility disorders include reduced sperm motility and quality, oxidative stress, reduced antioxidant capacity, mtDNA fragmentation, and sperm mitochondrial dysfunction.

Sperm contain a number of mitochondria that are spirally arranged around the middle part of the axomen. The main role of mitochondria in spermatozoa is to generate the energy needed for their motility (1, 2). Endogenous sources - coenzyme Q10 and carnitine - are key for energy production (ATP) in sperm mitochondria. Physiological functions of sperm require a minimal amount of reactive oxygen species (ROS), but uncontrolled ROS production contributes to reduced motility and sperm count, fragmentation of mtDNA (3).

In recent years, blood cells (platelets, lymphocytes and monocytes) have been used to diagnose mitochondrial disorders. Isolated peripheral blood platelets are an available source of mitochondria to assess mitochondrial health. Platelets receive energy mainly through glycolysis and oxidative phosphorylation. Platelet mitochondrial dysfunction has been demonstrated in patients with chronic kidney disease (4, 5), in patients with rheumatoid arthritis (6), in patients with acute COVID-19 (7). An O2k-respirometer (Oroboros, Austria) (8, 9) is used for respirometric analysis of platelet mitochondrial bioenergetics.

None information is available on the effect of infertility on platelet mitochondrial function, none on the effect of SARS-CoV-2 on platelet mitochondrial function in infertile patients, or the effect of vaccination on sperm function. Testicular damage and subsequent infertility due to SARS-CoV infection is expected. -2, directly via SARS-CoV-2 binding to ACE2 receptors or secondarily, in relation to the immunological and inflammatory response (10). SARS-CoV-2 virus induces excessive production of pro-inflammatory cytokines, mainly interleukin 6 (IL6), interleukin-1β (IL-1β) and tumor necrosis factor α (TNFα). Cytokines can impair sperm movement and reduce sperm count. High levels of pro-inflammatory cytokines have been found in infertile men (with oligozoospermia, asthenozoospermia, teratozoospermia) (11).

SARS-CoV-2 virus can manipulate mitochondrial function in patients with post-COVID-19 syndrome, which may persist for a long time (12). In previous our study the investigators found modulation of platelet mitochondrial respiration, reduction ATP production via oxidative phosphorylation, reduces endogenous coenzyme Q10 production, reprogramming of cellular metabolism patients after 4-7 weeks overcoming acute COVID-19, SARS-CoV-2 (7). In another studies the investigators confirmed platelet mitochondrial bioenergetic deficiency, reduced endogenous coenzyme Q10 production in patients with post-COVID-19 syndrome, 3-6 months after overcoming COVID-19 (13, 14, 15). Results of this study contribute to the understanding of the pathobiochemical mechanisms of infertility on subcellular level and to verify the hypothesis that infertility and the effect of SARS-CoV-2 on infertility may affect platelet mitochondrial bioenergetics and endogenous coenzyme Q10 levels.

ELIGIBILITY:
Inclusion Criteria:

* Infertile patients without COVID-19
* Infertile patients after COVID-19 Control group: healthy volunteers

Exclusion Criteria:

* disagreement with informed consent

Ages: 18 Years to 40 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Only men have sperm.
Enrollment: 45 (Actual)
Dates: Start 2022-04-01 (Actual); Primary Completion 2022-12-31 (Estimated); Study Completion 2023-03-30 (Estimated)

PRIMARY OUTCOMES:
Clinical symptoms | 15 minutes
  Clinical symptoms: infertile patients without COVID-19 (vaccinated, or none vaccinated) Clinical symptoms patients after COVID-19
Damaged platelet mitochondrial bioenergetics 1 | 1 day
  Basal oxygen consumption rate in intact platelets (ce)
Damaged platelet mitochondrial bioenergetics 2 | 1 day
  rate of mitochondria LEAK respiration with CI-linked substrates (1PM - state 4)
Damaged platelet mitochondrial bioenergetics 3 | 1 day
  CI-linked respiration coupled with ATPproduction (2D-CI-linked oxidative phosphorylation capacity), respiration after addition of cytochrome c (2C).
Damaged platelet mitochondrial bioenergetics 4 | 1 day
  Maximal oxidative capacity (the electron transfer capacity -ET), after uncoupler titration (3U).
Damaged platelet mitochondrial bioenergetics 5 | 1 day
  After addition of exogenous substrate glutamate (4G) non-coupled mitochondrial oxygen consumption.
Damaged platelet mitochondrial bioenergetics 6 | 1 day
  Non-coupled oxygen consumption with CI&CII-linked substrate (5S) improvement of mitochondrial parameters representing OXPHOS- and electron tranport capacity (ET-capacity).
Endogenous coenzyme Q10-TOTAL 1 | 1 day
  CoQ10-TOTAL in: Platelets (pmol.10-9 cells)
Endogenous coenzyme Q10-TOTAL 2 | 1 day
  CoQ10-TOTAL in: Blood (µmol.L-1)
Endogenous coenzyme Q10-TOTAL 3 | 1 day
  CoQ10-TOTAL in: Plasma (µmol.L-1)
Endogenous coenzyme TBARS | 1 day
  Endogenous concentration of CoQ10-TOTAL (ubiquinone + ubiquinol) in platelets, blood and plasma CoQ10-TOTAL in: TBARS in plasma (µmol.L-1).
Sperm analysis 1 | 1 day
  standard spermiogram examination (volume, pH, number, motility and pathology) in the broker chamber
Sperm analysis 2 | 1 day
  mioxsys for redox potential
Sperm analysis 3 | 1 day
  Vitalsperm (eosin-nigrosine staining) for sperm vitality
Sperm analysis 4 | 1 day
  anti-sperm antibody (IgG) test

CONTACTS AND LOCATIONS:
Overall Officials: Anna Gvozdjáková, Prof.Dr.DSc., Principal Investigator — CU in Bratislava, Faculty of Medicine, Pharmacobiochemical Laboratory of 3rd department of Medicine
Locations (1):
- Pharmacobiochemical Laboratory of Third Department of Internal Medicine, Faculty of Medicine Comenius University in Bratislava, Bratislava, Slovakia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Sheweita SA, Tilmisany AM, Al-Sawaf H. Mechanisms of male infertility: role of antioxidants. Curr Drug Metab. 2005 Oct;6(5):495-501. doi: 10.2174/138920005774330594. PMID 16248841
- [Result] Gvozdjakova A, Kucharska J, Dubravicky J, Mojto V, Singh RB. Coenzyme Q(1)(0), alpha-tocopherol, and oxidative stress could be important metabolic biomarkers of male infertility. Dis Markers. 2015;2015:827941. doi: 10.1155/2015/827941. Epub 2015 Feb 25. PMID 25810566
- [Result] Gvozdjakova A, Sumbalova Z, Kucharska J, Chladekova A, Rausova Z, Vancova O, Komlosi M, Ulicna O, Mojto V. Platelet mitochondrial bioenergetic analysis in patients with nephropathies and non-communicable diseases: a new method. Bratisl Lek Listy. 2019;120(9):630-635. doi: 10.4149/BLL_2019_104. PMID 31475544
- [Result] Gvozdjakova A, Sumbalova Z, Kucharska J, Komlosi M, Rausova Z, Vancova O, Szamosova M, Mojto V. Platelet Mitochondrial Respiration, Endogenous Coenzyme Q10 and Oxidative Stress in Patients with Chronic Kidney Disease. Diagnostics (Basel). 2020 Mar 23;10(3):176. doi: 10.3390/diagnostics10030176. PMID 32210203
- [Result] Gvozdjakova A, Sumbalova Z, Kucharska J, Szamosova M, Capova L, Rausova Z, Vancova O, Mojto V, Langsjoen P, Palacka P. Platelet mitochondrial respiration and coenzyme Q10 could be used as new diagnostic strategy for mitochondrial dysfunction in rheumatoid diseases. PLoS One. 2021 Sep 28;16(9):e0256135. doi: 10.1371/journal.pone.0256135. eCollection 2021. PMID 34582480
- [Result] Sumbalova Z, Kucharska J, Palacka P, Rausova Z, Langsjoen PH, Langsjoen AM, Gvozdjakova A. Platelet mitochondrial function and endogenous coenzyme Q10 levels are reduced in patients after COVID-19. Bratisl Lek Listy. 2022;123(1):9-15. doi: 10.4149/BLL_2022_002. PMID 34967652
- [Result] Pesta D, Gnaiger E. High-resolution respirometry: OXPHOS protocols for human cells and permeabilized fibers from small biopsies of human muscle. Methods Mol Biol. 2012;810:25-58. doi: 10.1007/978-1-61779-382-0_3. PMID 22057559
- [Result] Abobaker A, Raba AA. Does COVID-19 affect male fertility? World J Urol. 2021 Mar;39(3):975-976. doi: 10.1007/s00345-020-03208-w. Epub 2020 Apr 21. No abstract available. PMID 32318855
- [Result] Rajak P, Roy S, Dutta M, Podder S, Sarkar S, Ganguly A, Mandi M, Khatun S. Understanding the cross-talk between mediators of infertility and COVID-19. Reprod Biol. 2021 Dec;21(4):100559. doi: 10.1016/j.repbio.2021.100559. Epub 2021 Sep 1. PMID 34547545
- [Result] Gvozdjakova A, Klauco F, Kucharska J, Sumbalova Z. Is mitochondrial bioenergetics and coenzyme Q10 the target of a virus causing COVID-19? Bratisl Lek Listy. 2020;121(11):775-778. doi: 10.4149/BLL_2020_126. PMID 33164536
- [Result] Boguenet M, Bouet PE, Spiers A, Reynier P, May-Panloup P. Mitochondria: their role in spermatozoa and in male infertility. Hum Reprod Update. 2021 Jun 22;27(4):697-719. doi: 10.1093/humupd/dmab001. PMID 33555313
- [Result] Khalili MA, Leisegang K, Majzoub A, Finelli R, Panner Selvam MK, Henkel R, Mojgan M, Agarwal A. Male Fertility and the COVID-19 Pandemic: Systematic Review of the Literature. World J Mens Health. 2020 Oct;38(4):506-520. doi: 10.5534/wjmh.200134. Epub 2020 Aug 14. PMID 32814369